CLINICAL TRIAL: NCT03613181
Title: A Randomized Open-Label, Multi-Center Pivotal Study of ANG1005 Compared With Physician's Best Choice in HER2-Negative Breast Cancer Patients With Newly Diagnosed Leptomeningeal Carcinomatosis and Previously Treated Brain Metastases (ANGLeD)
Brief Title: ANG1005 in Leptomeningeal Disease From Breast Cancer
Acronym: ANGLeD
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Angiochem Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANG1005-CLN-07
Record Dates: First submitted 2018-07-17; First posted 2018-08-03 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2023-04

CONDITIONS: Leptomeningeal Carcinomatosis; Leptomeningeal Metastases; Brain Metastases; HER2-negative Breast Cancer
Keywords: ANG1005; Leptomeningeal carcinomatosis; Leptomeningeal disease; Leptomeningeal metastases; Brain metastases; HER2-negative; Breast cancer; Targeted therapy
MeSH Terms: conditions — Meningeal Carcinomatosis; Brain Neoplasms; Meningeal Neoplasms; Breast Neoplasms | interventions — paclitaxel-Angiopep-2 conjugate; Capecitabine; eribulin; Methotrexate

STUDY DESIGN:
Intervention Model Description: 1:1 randomization to experimental arm and comparator arm
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ANG1005 (Experimental): ANG1005 Investigational Drug
  Interventions: Drug: ANG1005
- Physician's Best Choice (Active Comparator): One of the protocol specified Physician's Best Choice therapies, assigned by the Investigator prior to randomization: capecitabine or eribulin or high-dose intravenous (IV) methotrexate.
  Interventions: Drug: Physician's Best Choice

INTERVENTIONS:
Drug: ANG1005 — Investigational drug
  Other Names: paclitaxel trevatide
  Arms: ANG1005
Drug: Physician's Best Choice — Active Comparator: one of 3 pre-determined choices of therapies: capecitabine or eribulin or high-dose IV methotrexate.
  Other Names: capecitabine; eribulin; high-dose IV methotrexate.
  Arms: Physician's Best Choice

SUMMARY:
This is an open-label Phase 3 study to see if ANG1005 can prolong survival compared to a Physician Best Choice control in HER2-negative breast cancer patients with newly diagnosed leptomeningeal disease and previously treated brain metastases.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years old
2. HER2-negative breast cancer
3. At least 2 months of expected survival
4. Newly diagnosed leptomeningeal carcinomatosis
5. Documented history of brain metastasis that has been previously treated with radiation therapy
6. Neurologically stable
7. Eastern Cooperative Oncology Group performance status grade ≤2
8. Adequate laboratory test results prior to first dose
9. Patients who are fertile must agree to remain abstinent or use reliable method of birth control

Exclusion Criteria:

1. Any prior treatment for leptomeningeal carcinomatosis, except emergency radiotherapy or shunt
2. Prior treatment with ANG1005
3. Patients who have not had radiotherapy for their brain metastases
4. Evidence of symptomatic intracranial hemorrhage or increased intracranial pressure
5. Patients for whom intrathecal therapy is the most appropriate therapy for leptomeningeal disease
6. Pregnancy or lactation and patients planning to be pregnant during the study
7. Peripheral neuropathy > Grade 2
8. Evidence of severe or uncontrolled diseases
9. Presence of an infection including abscess or fistulae, or known infection with hepatitis B or C or HIV
10. History of interstitial lung disease
11. Severe conduction disturbance
12. Central nervous system disease requiring immediate neurosurgical intervention
13. Known allergy to paclitaxel or any of its components
14. Contra-indication for contrast-enhanced MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Overall survival | From the date of randomization until death due to any cause, assessed for up to 2 years.

SECONDARY OUTCOMES:
Central nervous system progression-free survival | From the date of randomization until central nervous system progression, assessed for up to 2 years.
Central nervous system clinical benefit rate at 3, 6 and 12 months | At 3, 6 and 12 months.
6-month and 12-month overall survival rates | At 6 and 12 months.
Leptomeningeal carcinomatosis response rate | Assessed for up to 2 years from first patient randomised.
Duration of leptomeningeal carcinomatosis response | Assessed for up to 2 years from first patient randomised.
Overall survival in triple negative breast cancer patients | From the date of randomization until death due to any cause, assessed for up to 2 years.